CLINICAL TRIAL: NCT05045027
Title: Simultaneous Multinuclear (Na+/H+) Metabolic MRI in Brain Tumors
Brief Title: Simultaneous Multinuclear Metabolic MRI in Newly Diagnosed or Recurrent Glioma
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 21-000514; NCI-2021-08698 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-09-07; First posted 2021-09-16 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Glioma; Malignant Glioma; Recurrent Glioma; Recurrent Malignant Glioma
MeSH Terms: conditions — Glioma | interventions — X-Rays; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: AIM 1: Previous scan data from healthy subjects is collected and analyzed. AIM 2: Patients undergo MRI. Patients also undergo collection of tissue samples for IHC analysis.
  AIM 3: Patients undergo multinuclear metabolic imaging before and after immunotherapy and prior to surgical resection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Basic science (MRI, metabolic imaging, tissue collection) (Experimental): AIM 1: Previous scan data from healthy subjects is collected and analyzed.
  AIM 2: Patients undergo MRI. Patients also undergo collection of tissue samples for IHC analysis.
  AIM 3: Patients undergo multinuclear metabolic imaging before and after immunotherapy and prior to surgical resection.
  Interventions: Procedure: Biospecimen Collection; Procedure: Diagnostic Imaging; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of tissue samples
  Other Names: Biological Sample Collection
Procedure: Diagnostic Imaging — Undergo multinuclear metabolic imaging
  Other Names: Medical Imaging
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging

SUMMARY:
This clinical trial constructs and tests a novel multinuclear metabolic magnetic resonance imaging (MRI) sequence in patients with glioma (brain tumor) that is newly diagnosed or has come back (recurrent). This trial aims to develop new diagnostic imaging technology that may bridge gaps between early detection and diagnosis, prognosis, and treatment in brain cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Construct and test a novel multinuclear Na+-H+ metabolic MRI sequence with sensitivity to Sodium (Na+) concentration, Potential of Hydrogen (pH), and oxygen (O2).

II. Correlate Na+-, pH-, and O2-weighted MR image measurements with sodium-proton exchanger isoform-1 (NHE1) immunohistochemistry (IHC), bioenergetics, and gene expression using stereotactic image-guided biopsies from human brain tumors.

III. Quantify changes in Na+-, pH-, and O2-weighted MR images after neoadjuvant anti-PD-1 immunotherapy in recurrent glioblastoma (GBM) and explore associated changes in tumor biology.

OUTLINE:

AIM 1: Previous scan data from healthy subjects is collected and analyzed.

AIM 2: Patients undergo MRI. Patients also undergo collection of tissue samples for IHC analysis.

AIM 3: Patients undergo multinuclear metabolic imaging before and after immunotherapy and prior to surgical resection.

ELIGIBILITY:
Inclusion Criteria:

* AIM 1: Healthy volunteers with no evidence of brain tumors or neurologic disease
* AIM 1: Age 18+
* AIM 2: Newly diagnosed or recurrent suspected or confirmed glioma (low or high grade)
* AIM 2: 10 IDH mutant and 10 IDH wild type gliomas
* AIM 2: Clinically indicated for resective surgery or biopsy
* AIM 2: Age 18+
* AIM 2: Tumor size > 1x1x1 cm (measurable)
* AIM 3: Recurrent glioma enrolled in an immunotherapy trial or clinically indicated to receive immunotherapy including anti-PD1
* AIM 3: Age 18+

Exclusion Criteria:

* AIM 1: Cannot safely perform an MRI
* AIM 1: Age < 18
* AIM 2: Cannot safely perform an MRI or use of MRI contrast agents
* AIM 2: Age < 18
* AIM 3: Cannot safely perform an MRI or use of MRI contrast agents
* AIM 3: Age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-09-10 (Estimated); Study Completion 2027-09-10 (Estimated)

PRIMARY OUTCOMES:
Total sodium concentration | Up to 5 years
  Will calculate NaT using standard methodology and normalize it to ocular Na+ concentration, a constant 135 mmol/l. Will then test whether healthy tissue has a coefficient of variance (COV) of < 10% across all 20 subjects.
NHE1 expression | Up to 5 years
  Will create a comprehensive map of genes/pathways and unique cell subsets associated with NHE1 expression.
Tumor metabolism | Up to 5 years
  Will examine the correlation between baseline tumor metabolism and change in metabolism with respect to overall survival using Cox multivariable regression.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin M Ellingson, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States